CLINICAL TRIAL: NCT02836847
Title: A Multicentre, Open-label, Randomised, Controlled Study of Molecularly Precision Target Therapy Based on Tumor Molecular Profiling With GEMOX in Advanced or Recurrent Extrahepatic Cholangiocarcinoma and Gallbladder Carcinoma
Brief Title: Molecularly Target Therapy With GEMOX in Advanced or Recurrent Extrahepatic Cholangiocarcinoma and Gallbladder Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, liu yingbin, head of general surgery department，xin hua Hospital, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLY201507
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cholangiocarcinoma of the Extrahepatic Bile Duct; Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Cetuximab; Trastuzumab; Gefitinib; Lapatinib; Everolimus; Sorafenib; Crizotinib

ARMS (2):
- target therapy (Experimental): The patients wil receive conventional chemotherapy(GEMOX) combined with target agents according to the result of genomic and proteomic profiling of tumor tissue.
  Interventions: Procedure: biological test; Drug: GEMOX; Drug: Cetuximab; Drug: Trastuzumab; Drug: Gefitinib; Drug: Lapatinib; Drug: Everolimus; Drug: Sorafenib; Drug: Crizotinib
- GEMOX (Other): The patients wil receive conventional chemotherapy(GEMOX).
  Interventions: Procedure: biological test; Drug: GEMOX

INTERVENTIONS:
Procedure: biological test — mutation and signal pathway activation status analysis
Drug: GEMOX — Conventional chemotherapy:gemcitabine and oxaliplatin
Drug: Cetuximab
  Arms: target therapy
Drug: Trastuzumab
  Arms: target therapy
Drug: Gefitinib
  Arms: target therapy
Drug: Lapatinib
  Arms: target therapy
Drug: Everolimus
  Arms: target therapy
Drug: Sorafenib
  Arms: target therapy
Drug: Crizotinib
  Arms: target therapy

SUMMARY:
The purpose of this study is to evaluate the feasibility, efficacy and safety of target therapy according to genomic and proteomic profiling combined with GEMOX in advanced or recurrent extrahepatic cholangiocarcinoma and gallbladder carcinoma.

DETAILED DESCRIPTION:
Genomic profiling studies the deoxyribonucleic acid (DNA) of a tumor to detect genetic changes or abnormalities. immuno-histochemistry tests reveal the abnormal activation status of signal pathways involved in study.These information will be used to recommend target therapy which may be more likely to result in a beneficial response.Patients will receive target anti-tumor agents according to the result of genomic and proteomic profiling.

ELIGIBILITY:
Inclusion Criteria:

* Chinese；
* Stable vital signs, KPS≥60;
* Patients have a diagnosis of advanced or recurrent metastatic extrahepatic cholangiocarcinoma or gallbladder carcinoma by histopathology or cytopathology, who are not suitable for radical surgery or have progressed R1 resection or palliative surgery;
* Adequate fresh tumor tissue for genome sequencing and immuno-histochemistry test; harboring mutations or abnormal activation of erb-b2 receptor tyrosine kinase signal pathway components;
* At least one measurable and evaluable site of disease according to the RECIST criteria version 1.1;
* Life expectancy of more than 12 weeks;
* Adequate hepatic, hematologic and renal functions(ALT≤10×upper limit of normal (ULN), AST≤10×ULN, the Child-Pugh classification for class A or B, white blood cells≥3×10^9/L, neutrophils≥1.5×10^9/L, platelets≥80×10^9/L , hemoglobin ≥ 90g/L, creatinine clearance rate≥60ml/min;
* Volunteer for this study, have written informed consent and have good Patient compliance;
* Female patients of childbearing potential and their mates agree to avoid pregnancy.

Exclusion Criteria:

* Have received following treatment before this study:

  1. Anti-tumor molecular target therapy; anti-tumor chemotherapy in 6 months;
  2. lesions have been treated by irradiation;
  3. participate in other therapeutic or interventional clinical trials.
* Have central nervous system metastasis;
* History of other malignancies except carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and other malignancies for more than 5 years;
* Have symptomatic ascites and need for treatment;
* Have serious concurrent illness including, but not limited to

  1. uncontrolled congestive heart failure(NYHA classification grade III or IV), unstable angina pectoris, unstable cardiac arrhythmias, uncontrolled moderate or serious hypertension(systolic blood pressure >21.3 Kpa or diastolic blood pressure >13.3 Kpa);
  2. ongoing or active serious infection;
  3. uncontrolled diabetes mellitus;
  4. psychiatric illness which potentially hamper the ability to willingly give written informed consent and compliance with the study protocol;
  5. HIV infection;
  6. other serious illness considered not suitable for this study by investigators.
* be allergic or have contraindications to target medicines involved in this study, gemcitabine or oxaliplatin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 1 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year. The progression is defined consistent with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria for solid tumors.

SECONDARY OUTCOMES:
Overall survival | up to 2 years
Objective Response Rate | up to 1 year
  Objective Response Rate is defined as the percentage of patients with a complete or partial response to treatment, consistent with RECIST version 1.1 criteria for solid tumors.
Disease Control Rate | up to 1 year
  Disease Control Rate is defined as the percentage of patients with a complete or partial response to treatment or stable disease, consistent with RECIST version 1.1 criteria for solid tumors.
percentage of patients with Clinical Benefit Response | up to 1 year
  Composite measure based on patient-reported pain (per Faces pain scale revised), patient-reported pain medication, Karnofsky performance status(KPS), and weight. Clinical benefit is indicated by either:(a) improvement in pain (less pain intensity with stable or decreased pain medication; or less pain medication with stable or decreased pain intensity) with stable or improved KPS; or (b) improvement in KPS with stable or improved pain.With stable for KPS and pain, clinical benefit may be indicated with an observation of positive weight change.
  Clinical benefit response (CBR) was classified weekly and a patient was considered a clinical benefit responder if clinical benefit was observed and maintained over a 4 week period.

CONTACTS AND LOCATIONS:
Overall Officials: liu yingbin, PHD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided